CLINICAL TRIAL: NCT01682421
Title: Investigation of Treatment With Topical Corticosteroid After Posterior Lamellar Corneal Transplantation
Brief Title: Topical Steroid Treatment After Posterior Lamellar Corneal Transplantation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Anders Ivarsen, MD, PhD, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AUH_DSAEK_STEROID
Record Dates: First submitted 2012-09-04; First posted 2012-09-11 (Estimated); Last update posted 2014-05-02 (Estimated); Status verified 2014-04

CONDITIONS: Endothelial Dystrophy; Secondary Bullous Keratopathy; Posterior Lamellar Keratoplasty; Descemet's Stripping Endothelial Keratoplasty
MeSH Terms: interventions — Dexamethasone; methylacetylene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Weak steroid (Experimental): Initial treatment with dexamethasone 6x per day for two weeks, followed by Fluorometholone 4x per day for 2 months, 3x per day for 2 months, 2x per day for 2 months, and finally 1x per day continually during 2 years.
  Interventions: Drug: Weak steroid (Flurolon, Allergan)
- Potent steroid (Experimental): Initially Dexamethasone 6x per day for 2 weeks followed by 4x per day for one month, 3x per day for one month, 2x per day for one month, and finally 1x per day for one month - giving a total of 4,5 months of steroid treatment.
  Interventions: Drug: Potent steroid (Maxidex, Alcon)

INTERVENTIONS:
Drug: Weak steroid (Flurolon, Allergan)
  Other Names: Flurolon, Allergan
  Arms: Weak steroid
Drug: Potent steroid (Maxidex, Alcon)
  Other Names: Maxidex, Alcon
  Arms: Potent steroid

SUMMARY:
After corneal transplantation, topical corticosteroids are used to reduce the risk of rejection.

However, the optimal postoperative treatment regimen is unknown. In most cases, a topical steroid is administered for at least 6 months after surgery, but it remains to be determined whether potent steroids offer better protection than weak steroids. Also, the length of the treatment is debated.

Since the use of steroids is not without potential serious ocular side effects, it is of considerable importance to investigate these problems.

The study aims to examine the frequency of rejection episodes after posterior lamellar keratoplasty; specifically comparing a short course of potent steroids versus a long course of weak steroids.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated for primary or secondary corneal endothelial failure at the department of ophthalmology, Aarhus University Hospital

Exclusion Criteria:

* Not fulfilling the above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Freedom from rejection | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, Aarhus Universtity Hospital, Aarhus, Denmark